CLINICAL TRIAL: NCT00788489
Title: A Prospective Study to Evaluate the Role of 2-[18F]Fluoro-2-deoxy-D-glucose (FDG)-Positron Emission Tomography (PET), Breast Magnetic Resonance Imaging (MRI), and Breast Ultrasonography in Monitoring Tumour Responses in Patients With Locally Advanced Breast Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: A Prospective Study to Evaluate FDG-PET, Breast MRI, and Breast Ultrasonography in Monitoring Tumour Responses in Patients With Locally Advanced Breast Cancer (LABC) Undergoing Neoadjuvant Chemotherapy
Acronym: PETLAB
Status: Completed | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PETLAB-06Jan2006
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Locally Advanced Breast Cancer
Keywords: breast cancer; FDG-PET; MRI; chemotherapy; ultrasonography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall goal of this study is to determine how FDG-PET, breast MRI and breast ultrasound can be incorporated into the assessment of treatment responses in women with LABC undergoing neoadjuvant chemotherapy. A prospective cohort study will be conducted evaluating the ability of FDG-PET, breast MRI and breast ultrasound to detect the presence of residual tumour in patients with LABC who have completed treatment with neoadjuvant chemotherapy prior to mastectomy.

DETAILED DESCRIPTION:
Locally advanced breast cancer (LABC) is usually treated with neoadjuvant chemotherapy followed by surgery and radiation. At present, monitoring of tumour responses to chemotherapy is primarily carried out using physical examination at the beginning of each chemotherapy cycle. Differentiating viable tumour tissue from inflammation or fibrotic scar tissue can be difficult. There is a growing body of evidence that newer imaging techniques such as positron emission tomography (PET) and magnetic resonance imaging (MRI) may be better at determining whether or not the tumour is actually shrinking. The purpose of this study is to determine the sensitivity and specificity of PET, MRI and ultrasound in evaluating tumour responses to chemotherapy in patients with LABC and compare this with physical examination, which is the current standard of care.

Two of the objectives of this study are to 1) determine whether PET, MRI or ultrasound have a higher sensitivity/specificity than physical examination alone in determining which LABC patients achieve a complete pathologic response following neoadjuvant chemotherapy, and 2) to investigate whether these additional investigations might lead to changes in clinical management by identifying non-responders earlier than with physical examination alone.

A prospective cohort study design will be conducted. Patients with LABC who receive chemotherapy will undergo physical examination, PET, MRI, and ultrasound at baseline, midway, and at the completion of chemotherapy. Approximately 100 patients will be accrued over a 5-year period.

This study will give clinicians further insight into the usefulness of PET, MRI, and ultrasound in monitoring treatment responses in patients with LABC. This could potentially lead to changes in clinical management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of breast cancer (invasive ductal or lobular carcinoma - not breast sarcoma or lymphoma)
* Patients having a clinical diagnosis of locally advanced breast cancer (T3 or T4, or N2 according to TNM classification) including inflammatory breast cancer.
* Patients must be able to undergo neoadjuvant chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 sufficient to undergo chemotherapy

Exclusion Criteria:

* Previously treated cancer other than nonmelanotic skin cancer or carcinoma in situ of the cervix, unless disease-free for 5 years or greater.
* Evidence of metastatic disease (found on chest X-ray, liver ultrasound or bone scan).
* Previous chemotherapy or hormonal therapy for breast cancer.
* Active infection or other significant illnesses which could hamper their ability to tolerate chemotherapy
* Significant concurrent medical problems (e.g. uncontrolled diabetes, active cardiac disease, severe chronic obstructive pulmonary disease) making the patient unfit for surgery.
* Any condition that could interfere with their ability to provide informed consent such as dementia or severe cognitive impairment.
* Pregnant or lactating females (e.g. positive serum B-hCG pregnancy test).
* Unable to lie supine for imaging with PET.
* Inadequate hematologic, renal and liver function as measured by CBC (WBC < 4.0 x 109, Hb < 100 g/L, plt count < 100 x 109), and abnormal hepatic transaminases (AST, ALT, GGT, alkaline phosphatase > 2x normal), elevated total bilirubin, and elevated serum creatinine (Cr > 110 micromol/L).
* Any contraindication to undergoing MRI or PET.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 patients will be accrued over a 5-year period.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2006-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are the sensitivity and specificity of physical examination, ultrasound, breast MRI and PET in predicting which patients have achieved a complete pathologic response (pCR) prior to undergoing surgery. | 5 years

SECONDARY OUTCOMES:
Comparison of mean SUV uptake on FDG-PET for patients with pCR versus patients without pCR following neoadjuvant chemotherapy | 5 years
The size of the tumour measured by physical examination, breast ultrasound and MRI just prior to surgery will be compared to pathology tumour measurements found following mastectomy. | 5 years
Retrospective modelling to assess whether imaging test midway through chemotherapy affect management decisions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Som Mukherjee, MD MSc FRCP(C), Principal Investigator — Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada